CLINICAL TRIAL: NCT01392898
Title: The Effect of Liraglutide on Insulin-associated wEight GAiN in Patients With Type 2 Diabetes Mellitus (ELEGANT Trial)
Brief Title: Liraglutide and Insulin Therapy in Patients With Type 2 Diabetes
Acronym: ELEGANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lir-HJCJ-03
Record Dates: First submitted 2011-07-04; First posted 2011-07-13 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: liraglutide; insulin; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Liraglutide; Insulin

ARMS (2):
- liraglutide (Experimental)
  Interventions: Drug: liraglutide
- insulin (Active Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: liraglutide — liraglutide 1.8 mg q.d.
  Arms: liraglutide
Drug: Insulin — insulin dosed according titration scheme
  Arms: insulin

SUMMARY:
Insulin therapy is frequently needed to achieve adequate glycaemic control in type 2 diabetes. Although insulin is an effective treatment modality, this is often at the expense of significant weight gain. Weight gain is obviously undesirable in an already overweight population, but may also deter further optimization of insulin therapy. Large inter-individual differences exist in the level of weight gain after initiation of insulin therapy, but no clear predictive factors have prospectively been identified thus far.

Liraglutide (Victoza®), a human glucagon-like peptide-1 (GLP-1) analogue, improves glycaemic control and reduces weight. We hypothesize that in patients who show (excessive) weight gain after introducing insulin therapy, adding liraglutide is effective in reversing body weight while preserving glycaemic control.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus on short-term (≤ 12 months) insulin therapy with concomitant documented weight gain of ≥ 4 % body weight will be selected and treated with liraglutide 1.8 mg sc q.d. for 26 weeks and compared to patients receiving standard care (continuation of insulin therapy without liraglutide) in an open-label, randomized study. After 26 weeks, patients receiving standard care will subsequently be treated with liraglutide for 26 weeks. The group on active liraglutide treatment will continue for an additional 26 weeks. In this way all patients can benefit from liraglutide.

All subjects will continue insulin therapy and oral hypoglycaemic agents (SU derivatives and metformin allowed) treatment. With respect to safety in order to avoid hypoglycaemic events, total insulin dose will be decreased by 20% when starting liraglutide. Within the first weeks after start of study medication patients will perform frequently self-measured capillary blood glucose profiles and will be instructed to adjust insulin dose if necessary. Initially, insulin dose will be adjusted weekly by telephone consultation. Thereafter, patients will perform blood glucose profiles prior to every outpatient visit. A liraglutide-insulin titration algorithm will be used to adjust insulin dose. Every 4-6 weeks patients will visit the hospital to assess body weight, to adjust insulin dose and to check for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus on short-term insulin therapy (≤ 12 months); all types of insulin allowed
* Documented insulin-associated weight gain ≥ 3.0 kg from the start of insulin therapy until inclusion
* Age 18-75 years
* BMI ≥ 25 kg/m2
* Stable glycaemic control mirrored by HbA1c ≥ 6.5 and ≤ 8.5 %

Exclusion Criteria:

* Inability to provide informed consent
* Type 1 diabetes mellitus, MODY diabetes, or LADA diabetes (presence of anti-GAD)
* Presence of any medical condition that might interfere with the current study protocol.
* Inflammatory bowel disease (e.g. M. Crohn, ulcerative colitis)
* Recurrent hypoglycaemic events
* Diabetic gastroparesis
* Heart failure (LVEF ≤ 30%)
* Use of TZDs (glitazones), DDP-IV (dipeptidylpeptidase-inhibitor)
* Use of medication associated with impaired glucose metabolism including corticosteroids
* Pregnancy or breast-feeding (contraception of at least 3 months before inclusion is required for fertile women)
* Pre-existing thyroid disease
* Liver disease (aspartate aminotransferase or alanine aminotransferase level of more than three times the upper limit of normal range)
* Renal disease (creatinine > 130 µmol/l or MDRD-GFR <30 ml/min/1.73m2)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Body weight change (measured body weight at 26 weeks minus baseline body weight) | 26 weeks (26 weeks - baseline)
  Measuring body weight after 26 weeks minus baseline body weight as the change in body weight after Liraglutide treatment.

SECONDARY OUTCOMES:
Measuring change in insulin dose (insulin dose at 26 weeks minus insulin dose at baseline) | 26 weeks (26 weeks -baseline)
  Change in insulin dose by measuring insulin dose at 26 weeks minus the insulin dose at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] de Wit HM, Vervoort GM, Jansen HJ, de Grauw WJ, de Galan BE, Tack CJ. Liraglutide reverses pronounced insulin-associated weight gain, improves glycaemic control and decreases insulin dose in patients with type 2 diabetes: a 26 week, randomised clinical trial (ELEGANT). Diabetologia. 2014 Sep;57(9):1812-9. doi: 10.1007/s00125-014-3302-0. Epub 2014 Jun 20. PMID 24947583